CLINICAL TRIAL: NCT03658954
Title: Development of a Multimodal Sleep Intervention Using Wearable Technology to Reduce Heavy Drinking in Young Adults
Brief Title: Multimodal Sleep Intervention Using Wearable Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000021048; R34AA026021 (NIH)
Record Dates: First submitted 2018-08-31; First posted 2018-09-06 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Drinking, Alcohol
Keywords: Sleep Disorders; Self-Management; Telemedicine; Health Education; Wearable Electronic Devices
MeSH Terms: conditions — Alcohol Drinking; Sleep Wake Disorders; Health Education | interventions — Counseling; Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: Random assignment to one of three groups in 2:1:1 ratio, each group receiving some variation on 2-week intervention. Measurements taken at baseline, 4 weeks, 8 weeks, 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Advice (Active Comparator): Participants receive only web-based sleep health advice
  Interventions: Behavioral: Advice
- Advice + Self-monitoring (Experimental): Participants receive web-based sleep health advice + sleep/alcohol smartphone diary self-monitoring
  Interventions: Behavioral: Advice; Behavioral: Self-monitoring
- Advice + Self-monitoring + Feedback (Experimental): Participants receive web-based sleep health advice + sleep/alcohol smartphone diary self-monitoring + 2 sessions of sleep/alcohol wearable/diary data feedback & tailored coaching
  Interventions: Behavioral: Advice; Behavioral: Self-monitoring; Behavioral: Feedback

INTERVENTIONS:
Behavioral: Advice — Once per week for two weeks, participants will come to in-person visits to receive brief web-based sleep health advice.
Behavioral: Self-monitoring — Participants will complete daily smartphone-based sleep and alcohol diaries for two weeks.
  Arms: Advice + Self-monitoring; Advice + Self-monitoring + Feedback
Behavioral: Feedback — Participants will receive feedback once per week for two weeks on their sleep and alcohol consumption, using all possible data derived from Philips actiwatches and SCRAM ankle biosensors & smartphone diaries & tailored coaching with a health coach
  Arms: Advice + Self-monitoring + Feedback

SUMMARY:
This research study is examining three different components of a digital sleep intervention: web-based sleep health advice, sleep and alcohol smartphone diary self-monitoring, and personalized sleep and alcohol consumption feedback from wearables/diaries and tailored coaching. The study is designed to find out which of these components are most effective for reducing alcohol use and improving sleep health among young adults. The study has three parts: 1) an intake session; 2) a 2-week treatment phase; and 3) three follow-up visits over the next 10 weeks.

DETAILED DESCRIPTION:
Targeting sleep concerns may be a novel strategy for reducing increased risk of alcohol use disorders in young adults. The current study will develop and test a multimodal digital intervention addressing sleep concerns in 120 heavy-drinking young adults. All participants will wear sleep and alcohol biosensors daily. Participants will be randomized to one of three interventions. The primary intervention (60 participants) will include web-based sleep health advice + sleep/alcohol smartphone diary self-monitoring + sleep/alcohol data wearable/diary feedback & tailored coaching. The comparison interventions will be compared to matched control conditions only including these components: (1) web-based sleep health advice (30 participants) or (2) web-based sleep health advice + sleep/alcohol smartphone diary self-monitoring (30 participants). The primary objective is to evaluate sleep intervention component feasibility, acceptability, and preliminary efficacy on alcohol and sleep outcomes to inform a large scale Stage II randomized trial comparing the final digital intervention against standard care for this population.

ELIGIBILITY:
Inclusion Criteria:

1. 18-25 years of age;
2. report ≥ 3 heavy drinking occasions in the last 2 weeks (i.e., ≥5 drinks on 1 occasion for men; ≥4 for women);
3. report having concerns about their sleep;
4. willing/able to complete daily smartphone diaries and wear sleep and alcohol trackers;
5. report Alcohol Use Disorders Identification Test - Consumption (AUDIT-C) scores indicative of risk of harm from drinking (i.e., ≥7 and ≥5 for men and women, respectively)
6. read and understand English;
7. have a smartphone

Exclusion Criteria:

1. history of a sleep disorder;
2. night or rotating shift work; travel beyond 2 time zones in month prior and/or planned travel beyond 2 time zones during study participation;
3. meet criteria for an alcohol use disorder in the past 12 months that is clinically severe defined by: a) a history of seizures, delirium, or hallucinations during alcohol withdrawal; b) report drinking to avoid withdrawal symptoms or have had prior treatment of alcohol withdrawal; c) have required medical treatment of alcohol withdrawal in the past 6 months;
4. currently enrolled in alcohol or sleep treatment;
5. exhibit current severe psychiatric illness (i.e., bipolar disorder, schizophrenia, major depression, panic disorder, organic mood or mental disorders, or suicide or violence risk) by history or psychological examination;
6. current DSM-V substance use disorder (other than cannabis) or a positive urine drug screen for opiates, cocaine, barbiturates, benzodiazepines, amphetamines, or phencyclidine.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fucito LM, Ash GI, Wu R, Pittman B, Barnett NP, Li CR, Redeker NS, O'Malley SS, DeMartini KS. Wearable Intervention for Alcohol Use Risk and Sleep in Young Adults: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2513167. doi: 10.1001/jamanetworkopen.2025.13167. PMID 40445615
- [Derived] Griffith FJ, Ash GI, Augustine M, Latimer L, Verne N, Redeker NS, O'Malley SS, DeMartini KS, Fucito LM. Natural language processing in mixed-methods evaluation of a digital sleep-alcohol intervention for young adults. NPJ Digit Med. 2024 Nov 29;7(1):342. doi: 10.1038/s41746-024-01321-3. PMID 39613828
- [Derived] Fucito LM, Ash GI, DeMartini KS, Pittman B, Barnett NP, Li CR, Redeker NS, O'Malley SS. A Multimodal Mobile Sleep Intervention for Young Adults Engaged in Risky Drinking: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Feb 26;10(2):e26557. doi: 10.2196/26557. PMID 33635276

RESULTS

PARTICIPANT FLOW:
Groups:
- Advice: Participants receive only web-based sleep hygiene advice
  Advice: Once per week for two weeks, participants will come to in-person visits to receive brief web-based sleep hygiene advice.
- Advice + Self-monitoring: Participants receive web-based sleep hygiene advice + sleep/alcohol diary self-monitoring
  Advice: Once per week for two weeks, participants will come to in-person visits to receive brief web-based sleep hygiene advice.
  Self-monitoring: Participants will complete daily web-based sleep and alcohol smartphone diaries for two weeks.
- Advice + Self-monitoring + Feedback: Participants receive web-based sleep hygiene advice + sleep/alcohol diary self-monitoring + sleep/alcohol data feedback
  Advice: Once per week for two weeks, participants will come to in-person visits to receive brief web-based sleep hygiene advice.
  Self-monitoring: Participants will complete daily web-based sleep and alcohol smartphone diaries for two weeks.
  Feedback: Participants will receive feedback once per week for two weeks on their sleep and alcohol consumption, using all possible data derived from Philips actigraphs and SCRAM blood-alcohol trackers and smartphone diary data.
Period: Overall Study
Arm/Group | Advice | Advice + Self-monitoring | Advice + Self-monitoring + Feedback
Started | 30 | 30 | 60
Completed 2 Week Treatment | 28 | 30 | 60
Completed 12 Week Follow-up | 27 | 29 | 59
Completed | 28 | 30 | 60
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 120 randomized participants that began the study.
Groups:
- Advice + Self-monitoring: Participants receive web-based sleep hygiene advice + sleep/alcohol diary self-monitoring
  Advice: Once per week for two weeks, participants will come to in-person visits to receive brief web-based sleep hygiene advice.
  Self-monitoring: Participants will complete daily web-based sleep and alcohol diaries for two weeks.
- Advice + Self-monitoring + Feedback: Participants receive web-based sleep hygiene advice + sleep/alcohol diary self-monitoring + sleep/alcohol data feedback
  Advice: Once per week for two weeks, participants will come to in-person visits to receive brief web-based sleep hygiene advice.
  Self-monitoring: Participants will complete daily web-based sleep and alcohol diaries for two weeks.
  Feedback: Participants will receive feedback once per week for two weeks on their sleep and alcohol consumption, using all possible data derived from Fitbit actigraphs and Milo Sensor blood-alcohol trackers.
- Total: Total of all reporting groups
Arm/Group | Advice | Advice + Self-monitoring | Advice + Self-monitoring + Feedback | Total
Number analyzed (Participants) | 30 | 30 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.9 (1.7) | 21.3 (1.8) | 21.2 (1.7) | 21.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 30 | 61
  Male | 15 | 14 | 30 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 9 | 19
  Not Hispanic or Latino | 25 | 25 | 51 | 101
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 7 | 9
  White | 26 | 25 | 45 | 96
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Total Alcohol Drinks Consumed Over the 12wk Followup
Description: This will be recorded using the Timeline Follow-back Interview, based on the U.S. Standard Drink Conversion Chart. Upon results entry, the outcome was updated to include the following: data are log-transformed total alcohol drinks consumed over time from Week 4 to Week 12 follow-up, controlling for baseline.
Time Frame: weeks 4 through 12
Population: Intention to treat analysis
Measure: Least Squares Mean (Standard Error); unit: log-transformed total alcohol drinks
Arm/Group | Advice | Advice + Self-monitoring | Advice + Self-monitoring + Feedback
Number analyzed (Participants) | 30 | 30 | 60
log-transformed total alcohol drinks | 3.07 (0.13) | 2.95 (0.12) | 2.96 (0.09)
Statistical Analysis 1: Comparison: Advice vs Advice + Self-monitoring vs Advice + Self-monitoring + Feedback; Testing for group effect; Test type: Superiority; p = 0.75, Mixed Models Analysis

2. Secondary Outcome: National Institutes of Health Patient-Reported Outcomes Measurement Information System™ (NIH PROMIS™) Sleep Disturbance Score- Least Squares Mean Across Assessments
Description: This is a validated, reliable measure of perceived sleep quality/satisfaction and difficulty initiating/maintaining sleep. Upon results entry, the outcome was updated to reflect the following: Sleep Disturbance Score assessed at Week 4, 8 and 12, controlling for baseline. Scores represent standardized T scores with mean of 50 and a standard deviation of 10. Higher scores, 50 and above, equal greater sleep disturbance. Scores 60 and above are clinically significant. Presented is the least squares mean across assessments.
Time Frame: Baseline, week 4, week 8 and week 12
Population: Intention to treat analysis
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Advice | Advice + Self-monitoring | Advice + Self-monitoring + Feedback
Number analyzed (Participants) | 30 | 30 | 60
T-score | 51.39 (0.67) | 49.75 (0.65) | 49.46 (0.45)
Statistical Analysis 1: Comparison: Advice vs Advice + Self-monitoring vs Advice + Self-monitoring + Feedback; Testing for group effect; Test type: Superiority; p = 0.05, Mixed Models Analysis

3. Secondary Outcome: National Institutes of Health Patient-Reported Outcomes Measurement Information System™ (NIH PROMIS™) Sleep-Related Impairment Score - Least Squares Mean Across Assessments
Description: National Institutes of Health Patient-Reported Outcomes Measurement Information System™ (NIH PROMIS™) Sleep-Related Impairment Score assessed at Week 4, 8, and 12, controlling for baseline. Scores represent standardized T scores with mean of 50 and a standard deviation of 10. Higher scores, 50 and above, equal greater sleep-related impairment. Scores 60 and above are clinically significant. Presented is the least squares mean across assessments.
Time Frame: Baseline, week 4, week 8 and week 12
Population: Intention to treat analysis
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Advice | Advice + Self-monitoring | Advice + Self-monitoring + Feedback
Number analyzed (Participants) | 30 | 30 | 60
T-score | 57.80 (0.90) | 57.05 (0.88) | 54.89 (0.62)
Statistical Analysis 1: Comparison: Advice vs Advice + Self-monitoring vs Advice + Self-monitoring + Feedback; Testing for group effect; Test type: Superiority; p = 0.02, Mixed Models Analysis

4. Secondary Outcome: End of Treatment Satisfaction Survey Score
Description: In this survey, participants will rate their satisfaction associated with each intervention component using a 5-point Likert-type scale. Upon results entry, the outcome was corrected to reflect the following: the overall treatment satisfaction uses the mean of questions on a 5-point Likert-type scale from 0 to 4, with higher scores indicating greater satisfaction.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Advice | Advice + Self-monitoring | Advice + Self-monitoring + Feedback
Number analyzed (Participants) | 29 | 29 | 60
score on a scale | 3.45 (0.74) | 3.48 (0.57) | 3.60 (0.56)

5. Other Pre Specified Outcome: Stop-signal Reaction Time
Description: The difference between the mean reaction time and the stop-signal delay on the stop-signal test. Upon results entry, the following was added: This outcome will be explored as a potential mechanism of sleep intervention condition effects on the primary outcome of total drinks consumed. If there is a significant effect of condition on total drinks, the analysis of stop signal reaction time will be conducted. Due to COVID-19, this assessment was stopped since it could not be administered virtually. Since there was no effect of condition on total drinks consumed, an analysis of this outcome as a potential mechanism was not undertaken. The following represents the number of participants in each condition had this assessment conducted prior to COVID.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Advice | Advice + Self-monitoring | Advice + Self-monitoring + Feedback
Number analyzed (Participants) | 30 | 30 | 60
Participants | 22 | 19 | 43

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Advice | Advice + Self-monitoring | Advice + Self-monitoring + Feedback
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/60
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT03658954/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT03658954/ICF_001.pdf